CLINICAL TRIAL: NCT05742230
Title: Effect of Henagliflozin on Cardiac Function in Type 2 Diabetes Patients With Chronic Heart Failure: a Multicenter, Prospective, Pragmatic Randomized Controlled Trial
Brief Title: Effect of Henagliflozin on Cardiac Function in Type 2 Diabetes Patients With Chronic Heart Failure (HERO-HF)
Acronym: HERO-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1049
Record Dates: First submitted 2023-02-15; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Henagliflozin
MeSH Terms: conditions — Heart Failure | interventions — henagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Henagliflozin 10 mg (Experimental): Single 10 mg tablet, administered orally once daily for 12 weeks
  Interventions: Drug: Henagliflozin 10 mg
- blank control (Other): standard treatment
  Interventions: Drug: blank control

INTERVENTIONS:
Drug: Henagliflozin 10 mg — Participants will receive 10 mg single oral tablets orally once daily.
  Arms: Henagliflozin 10 mg
Drug: blank control — standard treatment
  Arms: blank control

SUMMARY:
The purpose of this study is to determine the superiority of the effectiveness of Henagliflozin 10 milligram (mg) daily versus blank control in participants with type II diabetes (T2DM) and symptomatic heart failure (HF) in improving the overall Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Score (CSS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM aged ≥18 years
* 6.5%≤HbA1c≤11%
* Clinically stable symptomatic heart failure

  (a) For HFrEF: (a) Ejection fraction (EF) less than or equal to (<=) 40% and (b) diagnosis of chronic heart failure within the past 18 months (B) For HFpEF: (a) EF greater than (>) 40%; (b) Diagnosis of chronic heart failure within the past 18 months
* Symptoms of heart failure at visit 1 (NYHA II-IV)
* KCCQ-OSS score < 80 at screening visit
* NT-proBNP > 125 pg/mL, or NT proBNP > 365 pg/mL in atrial fibrillation patients; Or BNP > 35 pg/mL, or BNP > 105 pg/mL in atrial fibrillation patients at screening visit
* Subject must have received (and be receiving) at least one stable optimal dose of guidelines recommended HF drugs (e.g., ACEi, ARB, ARNI, beta blockers, oral diuretics, MRA) prior to visit 1
* eGFR≥30 ml/min/1.73m2 at screening visit (CKD-EPI formula)
* Signed and dated written ICF

Exclusion Criteria:

* Pregnant and lactating women and women of childbearing age who do not want to use reliable contraception
* Known allergy to Henagliflozin
* Hospitalization for acute coronary syndrome, percutaneous coronary intervention, or cardiac surgery within 4 weeks before the screening visit
* Acute decompensated heart failure or hospitalization for decompensated heart failure within 4 weeks
* History of heart transplantation or ventricular assist device (VAD), or intention to heart transplantation or VAD
* Perinatal or chemotherapy-induced cardiomyopathy within 12 months
* Documented untreated ventricular arrhythmias with syncope within 3 months
* Diagnosed respiratory diseases
* Type I diabetes
* T2DM with history of ketoacidosis (DKA)
* Uncontrolled hypertension, defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg at screening visit
* Symptomatic hypotension and/or systolic blood pressure <90 mmHg at visit 0 or visit 1, or hypovolemia
* History of recurrent urinary and reproductive tract infections
* Current use or prior use of a SGLT-2i or GLP-1RA within 3 months
* Diagnosed malignant tumors
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1932 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Kansas City Cardiomyopathy Questionnaire-Clinical Summary Score (KCCQ-CSS) at Week 12 | 12 weeks
  Change from baseline in KCCQ-TSS was reported. KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. KCCQ-CSS is defined as the mean of the following available summary scores: Physical Limitation Score and Total Symptom Score.

SECONDARY OUTCOMES:
Change From Baseline in Kansas City Cardiomyopathy Questionnaire-Clinical Summary Score (KCCQ-CSS) at Week 4 | 4 weeks
  Change from baseline in KCCQ-TSS was reported. KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. KCCQ-CSS is defined as the mean of the following available summary scores: Physical Limitation Score and Total Symptom Score.
Change From Baseline in Kansas City Cardiomyopathy Questionnaire-Total Symptom Score (KCCQ-TSS) at Week 4, 12 | 4 weeks, 12 weeks
  KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. KCCQ-TSS was average of domains- symptom frequency and symptom burden.
Change From Baseline in NT-proBNP or BNP at Week 4, 12 | 4 weeks, 12 weeks
Change From Baseline in LV ejection fraction at Week 4, 12 | 4 weeks, 12 weeks
Change From Baseline in E/e' at Week 4, 12 | 4 weeks, 12 weeks
Change From Baseline in UACR at Week 4, 12 | 4 weeks, 12 weeks
Change From Baseline in eGFR at Week 4, 12 | 4 weeks, 12 weeks
Change From Baseline in HbA1c at Week 12 | 12 weeks
Change From Baseline in body weight at Week 4, 12 | 4 weeks, 12 weeks
Change From Baseline in BMI at Week 4, 12 | 4 weeks, 12 weeks
Change From Baseline in waist circumference at Week 4, 12 | 4 weeks, 12 weeks
Change From Baseline in lipids at Week 4, 12 | 4 weeks, 12 weeks
Change From Baseline in blood pressure at Week 4, 12 | 4 weeks, 12 weeks

OTHER OUTCOMES:
Occurrence of aggravated heart failure event | up to 12 weeks
Occurrence of cardiovascular (CV) death | up to 12 weeks
Occurrence of major renal events | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, MD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China